CLINICAL TRIAL: NCT00901823
Title: A Randomized, Open-Label, Single- and Multiple-Dose, Four-Way Parallel Study Comparing the Fed and Fasted Pharmacokinetics of Two Dose Levels of Diazoxide Choline Controlled-Release Tablet (DCCR) in Healthy VolunteersVOLUNTEERS
Brief Title: Open-Label, Single- and Multiple-Dose Pharmacokinetic Study of Diazoxide Choline
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not support the planned development of DCCR in the new indication
Sponsor: Essentialis, Inc. (Industry)
Responsible Party: Neil M Cowen, PhD/Chief Scientific Officer, Essentialis Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK010
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Single dose of low dose DCCR followed by a 14 day washout, then re-randomized to either low or high multiple dose DCCR
  Interventions: Drug: Diazoxide choline
- Sequence 2 (Experimental): Single dose of high dose DCCR followed by a 14 day washout, then re-randomized to either low or high multiple dose DCCR
  Interventions: Drug: Diazoxide choline high dose

INTERVENTIONS:
Drug: Diazoxide choline — A single dose low dose DCCR then re-randomized to either multiple dose low dose DCCR or high dose DCCR
  Arms: Sequence 1
Drug: Diazoxide choline high dose — A single dose high dose DCCR then re-randomized to either low or high multiple doses of DCCR
  Arms: Sequence 2

SUMMARY:
This is a single-center, randomized, open-label, single- and multiple-dose, five-treatment, two-period, four-way parallel study comparing the pharmacokinetics (PK) of Diazoxide Choline Controlled-Release Tablet (DCCR) administered orally under fed and fasting conditions at two dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy adults
* Fasting glucose ≤ 125 mg/dL and HbA1C ≤ 6.5
* Fasting triglyceride ≥150 mg/dL and ≤ 500 mg/dL

Exclusion Criteria:

* Known CAD, DM, uncontrolled HTN
* Pregnancy or unable to complaint with the birth control method required

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Compare the single-dose and steady-state, fed and fasting PK profiles of two dose levels of diazoxide administered as DCCR | 35 days

SECONDARY OUTCOMES:
Assess the impact of dosing in the absence of food on the steady-state pharmacokinetic profiles of two dose levels of diazoxide administered orally as DCCR under fed conditions | 35 days